CLINICAL TRIAL: NCT07230366
Title: Clinical Validation of AI-powered Smart Vehicle Assisted Gait Training in Neurodegenerative Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N202510104
Record Dates: First submitted 2025-10-02; First posted 2025-11-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease (PD); Dementia
Keywords: Neurodegenerative Diseases, Smart Electric Vehicles, Gait Training
MeSH Terms: conditions — Parkinson Disease; Dementia; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Gait abnormalities in patients with neurodegenerative diseases
  Interventions: Device: BestShape Go Intelligent Generation Transformable Electric Vehicle

INTERVENTIONS:
Device: BestShape Go Intelligent Generation Transformable Electric Vehicle — The specific applications of artificial intelligence in intelligent electric vehicles mainly include gait monitoring and analysis, real-time feedback and guidance, autonomous adaptive assistance, safety prevention and warnings, data collection and longterm tracking, as well as adding interactive and entertainment elements.

SUMMARY:
This study aims to verify the safety and preliminary clinical benefits of long-term gait training using AI-powered smart electric vehicles for patients with neurodegenerative diseases such as Parkinson's disease and dementia.

DETAILED DESCRIPTION:
This study is a single-center, prospective, open-label clinical intervention trial aimed at verifying the clinical safety and preliminary efficacy of an AI-powered smart electric vehicle in gait training for patients with Parkinson's disease and dementia. It is expected to recruit 120 participants aged 50-85 years, who will be randomly assigned to different training durations (2~12 weeks), with training sessions conducted two or three times a week, each lasting 30 to 60 minutes. The primary assessment indicators include gait speed, number of falls, and gait confidence scale, while secondary assessments include satisfaction and balance function. All study data will be coded and preserved for 10 years. The study is funded by the "Healthy Taiwan Cultivation Plan."

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neurodegenerative diseases (such as Parkinson's disease or dementia).
2. Age between 50-85 years.
3. Capable of walking for at least 10 meters, but may have unsteady gait or history of falls.
4. Able to understand the trial procedures and give informed consent.

Exclusion Criteria:

1. Severe cardiopulmonary disease or recent major surgery.
2. Unable to walk or requiring comprehensive physical support.
3. Severe cognitive impairment preventing understanding of the trial procedures or giving informed consent.
4. Visual or auditory impairments severe enough to prevent following trial instructions.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-12-10 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Before & after training (the training sessions will last for 2~12 weeks).

SECONDARY OUTCOMES:
Gait length | Before & after training (the training sessions will last for 2~12 weeks).
Number of falls | During 2~12 training sessions.
Patients' gait confidence scale | Before & after training (the training sessions will last for 2~12 weeks).
Patients' balance function | Before & after training (the training sessions will last for 2~12 weeks).
  Timed-up-and-Go Test
Patients' feedback | Before & after training (the training sessions will last for 2~12 weeks).
  Clinical Global Impression (CGI)

CONTACTS AND LOCATIONS:
Overall Officials: Lung Chan, MD, PhD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan